CLINICAL TRIAL: NCT04771416
Title: A Phase 1/2 Open-Label, Multicenter Dose-Ranging and Confirmatory Study to Assess the Safety, Tolerability and Efficacy of PBKR03 Administered to Pediatric Subjects With Early Infantile Krabbe Disease (Globoid Cell Leukodystrophy)
Brief Title: Study of Safety, Tolerability and Efficacy of PBKR03 in Pediatric Subjects With Early Infantile Krabbe Disease
Acronym: GALax-C
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to changes in the company strategy.
Sponsor: Gemma Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PBKR03-001; 2020-005229-95 (EudraCT Number)
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Leukodystrophy, Globoid Cell
Keywords: infantile; early infantile; Krabbe Disease; Rare disease; Leukodystrophy; GALC; Lysosomal storage disease
MeSH Terms: conditions — Leukodystrophy, Globoid Cell; Rare Diseases; Lysosomal Storage Diseases

STUDY DESIGN:
Intervention Model Description: Open-label, multi-center, dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation Cohorts designed to identify the optimal dose of PBKR03 (Experimental): Cohort 1: Subjects aged >4 to <9 months Drug: PBKR03 1.5 x 10^11 GC/g* Single dose of PBKR03, via intra cisterna magna
  Cohort 2: Subjects aged >4 to <9 months Drug: PBKR03 5.0 x 10^11 GC/g* Single dose of PBKR03, via intra cisterna magna
  Cohort 3: Subjects aged >1 to <4 months Drug: PBKR03 1.5 x 10^11 GC/g* Single dose of PBKR03, via intra cisterna magna
  Cohort 4: Subjects aged >1 to <4 months Drug: PBKR03 5.0 x 10^11 GC/g* Single dose of PBKR03, via intra cisterna magna
  *GC/g: genome copiesy per gram of estimated brain weight
  Interventions: Biological: PBKR03
- Part 2: Expansion Cohort designed to confirm the safety and efficacy of PBKR03 (Experimental): Cohort 5: Subjects aged >1 to <9 months Drug: PBKR03 Single dose of PBKR03, via intra cisterna magna Dose to be used for the confirmatory cohorts in Part 2 will be defined after a review of data from Part 1.
  *GC/g: genome copiesy per gram of estimated brain weight
  Interventions: Biological: PBKR03

INTERVENTIONS:
Biological: PBKR03 — Single dose of PBKR03, via intra cisterna magna

SUMMARY:
PBKR03 is a gene therapy for Krabbe Disease (Globoid cell leukodystrophy) intended to deliver a functional copy of the GALC gene to the brain and peripheral tissues. This study will evaluate the safety, tolerability and efficacy of this treatment by first evaluating two different doses in two different age groups, then confirming the optimal dose to be used for confirmation of safety and efficacy.

DETAILED DESCRIPTION:
PBKR03 is an adeno-associated viral vector serotype Hu68 carrying the gene encoding for human galactosylceramidase, GALC, formulated as a solution for injection into the cisterna magna.

This is a global interventional, multicenter, single-arm, dose escalation, study of PBKR03 delivered as a one-time dose administered into the cisterna magna of subjects with early infantile Krabbe Disease.

The dose-ranging portion of the study will enroll independent dose escalation cohorts in two age groups of subjects with early infantile Krabbe disease:

* Cohort 1: 3 subjects aged ≥4 to <9 months will receive the low dose (Dose I)
* Cohort 2: 3 subjects aged ≥4 to <9 months will receive the high dose (Dose II)
* Cohort 3: 3 subjects aged ≥1 to <4 months will receive the low dose (Dose I)
* Cohort 4: 3 subjects aged ≥1 to <4 months will receive the high dose (Dose II)

Part 1 of the study will enroll a total of four cohorts, enrolled sequentially with separate age-based dose-escalation cohorts. Enrollment will initiate in Cohort 1. Following completion of Cohort 1, simultaneous enrollment in Cohort 2 and Cohort 3 will occur. Cohort 4 will follow completion of cohort 3.

The confirmatory cohort, Part 2, will enroll subjects with early infantile Krabbe Disease, aged >1 to <9 months. These subjects will receive a dose chosen based on the data obtained in part 1 of the study This will be a 2-year study with a 3-year safety extension.

ELIGIBILITY:
Inclusion Criteria:

1. > 1 month and < 9 months of age at enrollment, either presymptomatic or symptomatic with first symptoms of Krabbe Disease at < 6 months of age
2. Leukocyte GALC activity below lower limit of normal (LLN)
3. Whole blood psychosine > 10 nM
4. Biallelic pathogenic GALC gene variants previously associated with early infantile Krabbe Disease or variants classified as likely pathogenic
5. Parents or the subject's legally authorized representative provide written informed consent prior to any study-related procedures, including screening evaluations
6. Symptomatic subjects must exhibit a minimum level of neurological and developmental function that indicates that they have the potential to benefit from treatment, at least with slowing or stabilization of their disease. In particular, the subject must demonstrate the following clinical features (when age-appropriate):

   * Thrusting of legs in play
   * Lifting of head
   * Eyes follow moving person
   * Smiles in response to speaker's attention

Exclusion Criteria:

1. Any clinically significant neurocognitive deficit not attributable to Krabbe disease.
2. An acute illness requiring hospitalization within 30 days of enrollment.
3. History of chronic ventilation assisted respiratory support (defined as more than 12 hours/day of bilevel positive airway pressure, continuous positive airway pressure (CPAP) or ventilator) or a need for tracheostomy as a result of their disease. Note: This does not exclude patients who use respiratory vests.
4. Intractable seizure or uncontrolled epilepsy defined as having had an episode of status epilepticus, or seizures requiring hospitalization.
5. Family history of seizures or epilepsy of infantile or childhood onset, other than febrile seizures. This does not exclude subjects with a family history of Krabbe disease.
6. Any contraindication to the ICM administration procedure, including contraindications to fluoroscopic imaging, intrathecal contrast and anesthesia or any condition that would increase the risk of adverse outcomes from the ICM procedure including, but not limited to, the presence of a space occupying lesion, aberrant vascular anatomy or congenital anatomical abnormalities such as a Chiari malformation.
7. Any contraindication to MRI or lumbar puncture (LP).
8. Prior gene therapy.
9. Enrollment in any other clinical study with an investigational product within 4 weeks prior to Screening or within 5 half-lives of the investigational product used in that clinical study, whichever is longer.
10. Prior Hematopoietic Stem Cell Transplantation (HSCT)
11. Receipt of a vaccine within 14 days prior to or after dosing.
12. Estimated glomerular filtration rate (eGFR) <60 mL/minute/1.73 m2 based on creatinine
13. Hematological abnormalities

    * Coagulopathy (INR > 1.5) or activated partial thromboplastin time [aPTT] > 40 seconds
    * WBC < 5.5 x 103 cells/ μL
    * Hemoglobin <10 g/dL
    * Thromobcytopenia (platelet count < 100,000 per μL.)
14. AST or ALT > 3 times the upper limit of normal (ULN) or total bilirubin > 1.5x ULN
15. Abnormal respiratory function

    1. Required suctioning in the absence of upper respiratory tract infection
    2. Hypoxemia (oxygen [O2] saturation awake less than 96% or O2 saturation asleep less than 96%, without ventilation support) as assessed during screening. Ventilatory support is defined as dependence on supplemental O2 or use of a ventilator or bilevel positive airway pressure (BiPap) or continuous positive airway pressure (Cpap) machine.
16. Poor peripheral perfusion or temperature instability in the absence of intercurrent illness
17. Medical conditions or laboratory or vital sign abnormalities that would increase risk of complications from intra-cisterna magna injection, anesthesia, fluoroscopy, LP, and/or MRI
18. Any condition (e.g., history of any disease, evidence of any current disease, any finding upon physical examination, or any laboratory abnormality) that, in the opinion of the investigator, would put the subject at undue risk during the administration procedure or would interfere with evaluation of PBKR01 or interpretation of subject safety or study results.

Ages: 1 Month to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs) and serious adverse events (SAEs) at Grade 3 or higher within 24 months of dosing | Up to 5 years (multiple visits)
  Assess the number of adverse events and serious adverse events at Grade 3 or higher as assessed by CTCAEv5.0
Change from baseline in nerve conduction and velocity in motor nerve conduction studies | From baseline to 5 years (multiple visits)
  NCS will measure velocity and amplitude in distal segments of the median, peroneal and tibial motor nerves to evaluate effects on peripheral nerve integrity.
Change from baseline in nerve conduction and velocity in sensory nerve conduction studies | From baseline to 5 years (multiple visits)
  NCS will measure velocity and amplitude in distal segments of the sural, radial and median sensory nerves to evaluate effects on peripheral nerve integrity
Number of Participants with Clinically Significant Laboratory Abnormalities as Measured Using Hematology, Chemistry and Coagulation Tests | Up to 5 years (multiple visits)
  Assess the number of participants with clinically significant laboratory changes including hematology, serum chemistry, and coagulation tests
Assess Humoral Response Against the Vector and Transgene in Serum | Up to 5 years (multiple visits)
  Assess serum antibody titers against AAVhu68 and against GALC following ICM administration of PBKR03
Assess Humoral Response Against the Vector and Transgene in CSF | Up to 5 years (multiple visits)
  Assess antibody titers in the cerebrospinal fluid against AAVhu68 and against GALC following ICM administration of PBKR03

SECONDARY OUTCOMES:
Change from Baseline in Developmental Milestones as Assessed by the Bayley Scale of Infant and Toddler Development, Third Edition | From baseline to 2 years (multiple visits)
  Assess changes in the developmental age and the total number of developmental milestones using the Bayley Scale of Infant and Toddler Development, Third Edition instrument
Change from Baseline in Developmental Milestones as Assessed by the Vineland Adaptive Behavior Scale-II | From baseline to 2 years (multiple visits)
  Assess changes in the developmental age and the total number of developmental milestones using the Vineland Adaptive Behavior Scale-II instrument
Change in Biomarkers of GALC Activity in Blood | From baseline to 2 years (multiple visits)
  Assess change in biomarkers of GALC activity in blood when compared with baseline
Change in Biomarkers of GALC Activity in CSF | From baseline to 2 years (multiple visits)
  Assess change in biomarkers of GALC activity when compared with baseline
Change in Biomarkers of GALC Substrates in Blood | From baseline to 2 years (multiple visits)
  Assess change in concentration of GALC substrates in blood
Change in Biomarkers of GALC Substrates in CSF | From baseline to 2 years (multiple visits)
  Assess change in concentration of GALC in CSF when compared with baseline
Change in Concentration of Biomarker of Disease Progression in Plasma | From baseline to 2 years (multiple visits)
  Assess change in neurofilament light chain (NfL) concentration as a marker for neurodegeneration and disease progression in plasma
Change in Concentration of Biomarker of Disease Progression in CSF | From baseline to 2 years (multiple visits)
  Assess change in neurofilament light chain concentration (NfL) as a marker for neurodegeneration and disease progression in CSF
Change in Brain Anatomy as Assessed by MRI | From baseline to 2 years (multiple visits)
  Assess change in disease severity, volumetric MRI measures, brain diffusivity, and white matter lesions by MRI imaging
Change in Quality of Life Using Pediatric Quality of Life Scale | From baseline to 2 years (multiple visits)
  Assess change in quality of life as measured by Pediatric Quality of Life Scale (Peds QL)
Change in Quality of Life Using Pediatric Quality of Life Scales | From baseline to 2 years (multiple visits)
  Assess change in quality of life as measured by the Pediatric Quality of Life - Infant Scale (PedsQL-IS)
Change in Ventilator-Free Survival Compared with Natural History Data | From baseline to 2 years (multiple visits)
  Assess change compared with natural history data in ventilator-free survival and chronic ventilatory support.
Incidence of Feeding Tube Placement at or Before Month 24 | 24 months
  Though speech and swallowing assessment, study participants will be evaluated to determine whether a feeding tube is warranted

CONTACTS AND LOCATIONS:
Overall Officials: May Orfali, MD, Study Director — Gemma Biotherapeutics
Locations (9):
- United States (4):
  - Ann & Robert Lurie, Chicago, Illinois
  - New York-Presbyterian, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah School of Medicine, Salt Lake City, Utah
- Hospital De Clinicas De Porto Alegre, Porto Alegre, Brazil
- Montreal Children's Hospital, Montreal, Canada
- Shaare Zadek Medical Center, Jerusalem, Israel
- Amsterdam UMC, Amsterdam, Netherlands
- Manchester University, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heller G, Bradbury AM, Sands MS, Bongarzone ER. Preclinical studies in Krabbe disease: A model for the investigation of novel combination therapies for lysosomal storage diseases. Mol Ther. 2023 Jan 4;31(1):7-23. doi: 10.1016/j.ymthe.2022.09.017. Epub 2022 Oct 4. PMID 36196048
- [Derived] Hordeaux J, Jeffrey BA, Jian J, Choudhury GR, Michalson K, Mitchell TW, Buza EL, Chichester J, Dyer C, Bagel J, Vite CH, Bradbury AM, Wilson JM. Efficacy and Safety of a Krabbe Disease Gene Therapy. Hum Gene Ther. 2022 May;33(9-10):499-517. doi: 10.1089/hum.2021.245. Epub 2022 Mar 22. PMID 35333110